CLINICAL TRIAL: NCT03627819
Title: The Effects of Plant Sterol and Plant Stanol Ester Enriched Foods on Biopsy Proven Liver Inflammation in NAFLD Patients - a Proof-of-concept Pilot Study
Brief Title: Plant Sterols and Plant Stanols and Liver Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry); Raisio Group (Industry); BASF (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH Pilot Study
Record Dates: First submitted 2018-07-18; First posted 2018-08-13 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Plant sterols; Plant stanols; Liver inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled, double blinded pilot study with a run-period of 2 weeks, an intervention period of 12 months and a wash-out period of 1 month.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The margarine is provided in white but colour-coded tubs and it is not known to the participant and the researcher which colour coded margarine is placebo, plant sterol or stanol ester margarine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Plant sterol-enriched margarine (Active Comparator): Intake of 20 gram margarine with added plant sterol esters, providing 3 gram plant sterols per day for 1 year
  Interventions: Dietary Supplement: Plant sterol-enriched margarine
- Plant stanol-enriched margarine (Active Comparator): Intake of 20 gram margarine with added plant stanol esters, 3 gram plant stanols per day for 1 year
  Interventions: Dietary Supplement: Plant stanol-enriched margarine
- Control margarine (Placebo Comparator): Intake of 20 gram margarine without any addition, every day for 1 year
  Interventions: Dietary Supplement: Control margarine

INTERVENTIONS:
Dietary Supplement: Plant sterol-enriched margarine — Margarine enriched with plant sterol esters
  Arms: Plant sterol-enriched margarine
Dietary Supplement: Plant stanol-enriched margarine — Margarine enriched with plant stanol esters
  Arms: Plant stanol-enriched margarine
Dietary Supplement: Control margarine — Margarine without any addition
  Arms: Control margarine

SUMMARY:
As the prevalence of obesity is reaching epidemic proportions, the prevalence of non-alcoholic fatty liver disease (NAFLD), including non-alcoholic steatohepatitis (NASH), increases concomitantly and becomes a major global health hazard. Successful pharmacological interventions to treat or prevent NASH are not available and so far only weight loss has clear benefits, but sustained weight-loss is difficult to achieve on the longer-term. We recently demonstrated in mice that plant sterol and stanol ester consumption inhibited the development of liver inflammation, which needs to be validated in humans in a translational approach. In the current proposed pilot study, the effect of consuming plant sterol or plant stanol esters on biopsy proven liver inflammation will be investigated in NAFLD patients.

The objective is to assess the effect of consuming plant sterol or plant stanol esters (3 grams/day) for 12 months on biopsy proven liver inflammation in NAFLD patients.

This study is a randomized, placebo-controlled, double blinded pilot study with a run-period of 2 weeks, an intervention period of 12 months and a wash-out period of 1 month.

The study population consists of 15 patients with biopsy-proven liver inflammation, aged 18-75 years.

All subjects will start a run-in period of two weeks during which they consume daily 20 grams of control margarine after which they will be randomly allocated to consume 20 grams control margarine or plant sterol or plant stanol enriched margarine on a daily basis for a period of 12 months. The primary outcome parameter in this study is biopsy proven liver inflammation.

DETAILED DESCRIPTION:
The objective is to assess the effect of consuming plant sterol or plant stanol esters (3 grams/day) for 12 months on biopsy proven liver inflammation in NAFLD patients.

This study is a randomized, placebo-controlled, double blinded pilot study with a run-period of 2 weeks, an intervention period of 12 months and a wash-out period of 1 month.

The study population consists of 15 patients with biopsy-proven liver inflammation, aged 18-75 years.

All subjects will start a run-in period of two weeks during which they consume daily 20 grams of control margarine after which they will be randomly allocated to consume 20 grams control margarine or plant sterol or plant stanol enriched margarine on a daily basis for a period of 12 months. The primary outcome parameter in this study is biopsy proven liver inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent
2. Diagnosed with liver inflammation by a liver biopsy <12 months prior to start of the study. All patients with biopsies older than 2 months must have a stable weight and biochemical liver test results. A certified, experienced pathologist will assess the presence of liver inflammation.
3. No presence of cirrhosis as diagnosed by the liver biopsy or by the FibroScan
4. Aged between 18 and 75 years
5. Body Mass Index (BMI) <40 kg/m2
6. Willingness to consume 20 grams of margarine on a daily basis for a period of 12 months

Exclusion Criteria:

1. Are less than 18 years of age or over 75 years of age
2. Females who are pregnant, breast feeding or who may wish to become pregnant during the study
3. Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, cancer or any condition which contraindicates, in the investigators judgement, entry to the study
4. Severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel disease and rheumatoid arthritis
5. Use of diuretics or insulin therapy
6. Use of anti-coagulants
7. History of illicit drug use
8. Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females
9. Not willing to stop the consumption of plant sterol or plant stanol enriched products 1 month before the start of the study (wash-in period)
10. Use of an investigational product in another biomedical study within the previous month
11. Contraindications for magnetic resonance imaging (MRI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Biopsy-proven liver inflammation | 1 year intervention
  NASH histology

SECONDARY OUTCOMES:
Hyperinsulinemic-euglycemic clamp | 1 year intervention
  Insulin sensitivity
Liver fat | 1 year intervention
  Liver fat measured by magnetic resonance spectroscopy (MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof., Study Chair — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No